CLINICAL TRIAL: NCT06283992
Title: Digital Health Navigation for Latino Patients With Type II Diabetes: A Randomized Controlled Trial
Brief Title: Digital Health Navigation for Latino Patients With Type II Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Jorge A. Rodriguez, MD, Assistant Professor, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2024p000095; K23MD016439 (NIH)
Record Dates: First submitted 2024-02-21; First posted 2024-02-28 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Type 2 Diabetes
Keywords: Latinos
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Researchers will compare effectiveness between two arms: 1) patient education using a digital navigator on using digital tools after discharge and 2) usual care (educational sheet).
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Digital Navigation (Experimental): Patients in this arm will receive 1:1 digital navigation support which will teach them about the functions of the patient portal and telehealth.
  Interventions: Other: Digital Navigation
- Standard of Care (No Intervention): Patients in this arm will receive the standard of care which will be an educational sheet.

INTERVENTIONS:
Other: Digital Navigation — 1:1 educational support at the bedside about the functions of the patient portal and telehealth that can help with care transitions.
  Arms: Digital Navigation

SUMMARY:
The goal of this clinical trial is to learn about digital literacy training in adult, Latino patient with type II diabetes. The main question it aims to answer is: Can providing digital literacy training during a hospital admission can help patients with their after-hospital care by using the patient portal and telehealth? Participants will receive digital literacy training by a digital navigator that focuses on the main patient portal functions. Researchers will compare patients who receive digital literacy training to those who receive standard of care (educational sheet) to see if it impacts their use of the patient portal after discharge.

DETAILED DESCRIPTION:
Latinos have the second-highest age-adjusted prevalence and among the highest incidence of diabetes. Latinos also experience worse glycemic control and diabetes-related complications, including diabetic retinopathy and chronic renal disease. These findings are concerning since Latinos are the largest minority group in the U.S and will account for 25% of the population by 2045.

Digital tools, like patient portals and telemedicine, offer an opportunity to address some of the challenges that lead to these disparities, especially during care transitions. However, Latinos, especially those who are Spanish-speaking are less likely to use digital health tools. Findings from previous health information technology work have highlighted barriers, including 1) digital access and literacy, 2) interface usability, 3) privacy, and 4) patient preference. One promising intervention to address digital literacy gaps is the use digital navigators.

This study aims are to assess a digital health navigation intervention focused on increasing patient portal use after discharge among Latino patients with type II diabetes admitted to the general medicine inpatient floor.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified Latino adult patients with type II diabetes
* Admitted to general medicine floors at Brigham and Women's Hospital
* Preferred language: English or Spanish

Exclusion Criteria:

* Critical illness
* dementia, delirium, or other condition that limits ability to participate in education and consent process

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2024-03-31 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants Who Login to the Portal | 30 days post-discharge
  Number of participants with at least 1 login to the portal in the 30 days after discharge

SECONDARY OUTCOMES:
Proportion of Participants that Perform Distinct Portal Functions | 30 days post-discharge
  Proportion of participants that perform distinct portal functions (sending messages, requesting refill)
Proportion of participants that complete a telehealth | 30 days post-discharge
  Proportion of participants that complete a telehealth visit during post-discharge period
Proportion of participants that are re-admitted | 30 days post-discharge
  Proportion of participants that are re-admitted within 30 days after discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided
There is no current plan to share data with other researchers.

REFERENCES:
- [Background] Rodriguez JA, Charles JP, Bates DW, Lyles C, Southworth B, Samal L. Digital healthcare equity in primary care: implementing an integrated digital health navigator. J Am Med Inform Assoc. 2023 Apr 19;30(5):965-970. doi: 10.1093/jamia/ocad015. PMID 36795062